CLINICAL TRIAL: NCT02654821
Title: Multicenter Phase I/IIa Study Using T-cell Receptor Gene Therapy in Metastatic Melanoma
Brief Title: Study With T-cel Receptor Gene Therapy in Metastatic Melanoma
Acronym: TCR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11TCR
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Stage IV Skin Melanoma; Eye; Melanoma
Keywords: Melanoma; TCR
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCR treatment (Experimental): Eligible patients will undergo leukapheresis to isolate autologous T cells. These T cells will be transduced with a retroviral vector encoding the 1D3 HM CysTCR, and subsequently expanded during short-term ex vivo culture. Following pre-treatment with nonmyeloablative chemotherapy, patients will receive the adoptive transfer of autologous, TCR transduced T cells.
  Interventions: Biological: TCR transduced T-cells; Procedure: Biopsy; Procedure: Blood taking

INTERVENTIONS:
Biological: TCR transduced T-cells — Eligible patients will undergo leukapheresis to isolate autologous T cells. These T cells will be transduced with a retroviral vector encoding the 1D3 HM CysTCR, and subsequently expanded during short-term ex vivo culture. Following pre-treatment with nonmyeloablative chemotherapy, patients will receive the adoptive transfer of autologous, TCR transduced T cells.
Procedure: Biopsy — During screening, after treatment and at time of regression/progression a biopsy will be taken for translational research.
Procedure: Blood taking — During screening, after the infusion with T-cells, after treatment and at time of regression/progression blood will be taken for translational research.

SUMMARY:
Patients with stage IV melanoma (also eye melanoma) will be treated with TCR transduced cells.

DETAILED DESCRIPTION:
In this multicenter phase I/IIa trial 25 patients will be treated with non-myeloablative chemotherapy followed by adoptive transfer of autologous TCR transduced T cells, to study the feasibility, safety and efficacy of this treatment.

Patients will receive a non-myeloablative lymphocyte-depleting preparative regimen consisting of cyclophosphamide (60 or 30 mg/kg/day x 2 days i.v.) and fludarabine (25 mg/m2/day i.v. x 5 days). Following this regimen, patients will receive one single intravenous adoptive transfer of transduced T cells starting with the first dose level.

* Dose level 1: 5x10^7 transduced T cells, cyclophosphamide 60 mg/kg/day
* Dose level 1a: 1,0x10^8 transduced T cells, cyclophosphamide 30 mg/kg/day
* Dose level 2: 2,5x10^8 transduced T cells, cyclophosphamide 60 mg/kg/day
* Dose level 3: maximum 1x10^9 transduced T cells (depending on production yield). At time points 4, 8, and 12 weeks and every 3 months thereafter patients will be evaluated for response to treatment. After 3 patients have been treated in each dose level, but not before 8 weeks after the last patient has been infused with transduced T cells, the DSMB will be informed about the observed toxicity and efficacy within this cohort and decide, based on this information, whether the trial will be continued to the next dose level or will continue in the current dose level. The study will continue as the first stage (2-stage Simon), until a total of 16 patients have been enrolled and treated: if less than 2 responses are observed, the trial will be stopped and the conclusion will be that TCR lacks efficacy. Otherwise, the trial will continue its second stage. In addition, safety data after these first 16 patients will be evaluated by the DSMB. Any unexpected or serious (grade 3/4 or higher) toxicities during the trial, will be reported immediately to the DSMB and CCMO. Second stage: overall 25 patients will be enrolled (including the first stage): if the total number of responses for the two stages combined is less than 5, the trial will be stopped as soon as this is evident and the conclusion will be that TCR lacks efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age.
* Patients must have inoperable stage IIIc or stage IV melanoma (AJCC), including ocular or mucosal melanoma, progressing after standard of care therapy, if available.
* Patients must be HLA-A*0201 positive.
* The primary tumor and/or metastasis have to be positive for MART-1 (>10% of tumor cells).
* Patients with measurable disease (RECIST 1.1)
* Patients must have a clinical performance status of ECOG 0 or 1.
* Patients of both genders must be willing to practice a highly effective method of birth control during treatment and for four months after receiving the preparative regimen.
* Patients must be able to understand and sign the Informed Consent document. Specific lab values

Exclusion Criteria:

* Life expectancy of less than three months.
* Requirement for systemic steroid therapy.
* Patients who have a history of CNS metastases.
* Patients with malignant pleural effusion or ascites.
* Any immunosuppressive chemotherapy or systemic steroid therapy within the last 3 weeks.
* Patients who have: history of coronary revascularization, documented LVEF of less than 45%, clinically significant atrial and/or ventricular arrhythmias including but not limited to atrial fibrillation, ventricular tachycardia, 2° or 3° heart block, documented FEV1 less than or equal to 60% predicted for patients with a history of cigarette smoking (greater than 20 pack/year within the past 2 years) and with symptoms of respiratory distress
* All patients' toxicities due to prior non-systemic treatment must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures or focal palliative radiotherapy (to non-target lesions) within the past 4 weeks, as long as all toxicities have recovered to grade 1 or less.
* Women who are pregnant or breastfeeding, because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. A negative pregnancy test before inclusion in the trial is required for all women of child bearing potential.
* Any active systemic infections, coagulation disorders or other active major medical illnesses, such as active autoimmune disease requiring anti-TNF treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the TCR treatment (according to CTCAE 4.0) | Baseline until release from the hospital, about 4 weeks.
  Safety of the TCR treatment will be measured by noting the toxicity (according to CTCAE 4.0) that the patient experiences while on treatment.
Objective response rate according to RECIST 1.1. | Baseline until progressive disease, median 6 months.
  The objective response rate will be measured by RECIST 1.1.

SECONDARY OUTCOMES:
1-year progression free survival (PFS) | Baseline until 1 year after treatment.
  1-year PFS will we measured by the number of patients still free of disease after 1 year, using RECIST 1.1 to measure progressive disease
Efficacy of induction of tumor specific T cell responses as measured by the persistence of Melan-A/MART1 specific T cells in peripheral blood samples | Baseline until progressive disease, median 6 months.
  Efficacy of induction of tumor specific T cell responses as measured by the persistence of Melan-A/MART1 specific T cells in peripheral blood samples at several time points following adoptive transfer and in tumor biopsies when possible.
Overall survival | Assessed up to 12 months
Systemic release of inflammatory cytokines after administration of transduced T cells compared to baseline | Baseline until progressive disease, median 6 months.
  To study whether the infusion of MART-1 specific TCR (1D3 HMCys) transduced T cells will lead to systemic release of inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: John B.A.G. Haanen, Prof., Principal Investigator — Antoni van Leeuwenhoek Ziekenhuis
Locations (1):
- Antoni van Leeuwenhoek ziekenhuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided